CLINICAL TRIAL: NCT06846619
Title: Patient Satisfaction of Intra-orally Scanned Versus Extra-orally Scanned Digitally Printed Maxillary Denture in Completely Edentulous Patients, in Vivo Study.
Brief Title: "Patient Satisfaction with Intra-Oral Vs. Extra-Oral Scanned 3D-Printed Dentures: an in Vivo Study"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lujayn Amr Mahmoud, Master Degree Student, Removable prosthodontics department, Faculty of Dentistry, CairoUniversity, Cairo University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12-2024
Record Dates: First submitted 2024-12-22; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Complete Edentulism
Keywords: Intraoral scanning; Extra oral scaning; Complete edentulism; Digital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-Orally Scanned Dentures (Experimental): Arm Description:
  Participants in this arm will receive maxillary dentures fabricated using intra-oral scanning technology. Digital impressions of the oral cavity will be captured directly using the 3Shape TRIOS intraoral scanner, eliminating the need for conventional impression materials. These digital impressions will be used to design and 3D-print the dentures, which will then be fitted and evaluated for comfort, fit, and aesthetics. Participants will wear these dentures for a specified period and provide feedback through structured satisfaction surveys.
  Interventions: Device: Intra-Oral Scanning Method; Device: Extra orally scanned
- Extra-Orally Scanned Dentures (Active Comparator): Arm Description:
  Participants in this arm will receive maxillary dentures fabricated using extra-oral scanning technology. Conventional impressions of the oral cavity will first be taken using traditional impression materials. These impressions will then be scanned externally using the 3Shape scanner to create digital models. The digital models will be used to design and 3D-print the dentures, which will then be fitted and evaluated for comfort, fit, and aesthetics. Participants will wear these dentures for a specified period and provide feedback through structured satisfaction surveys.
  Interventions: Device: Intra-Oral Scanning Method; Device: Extra orally scanned

INTERVENTIONS:
Device: Intra-Oral Scanning Method — Intervention Description:
  The intra-oral scanning method involves capturing digital impressions of the oral cavity directly using the 3Shape scanner. This method eliminates the need for traditional impression materials, providing a more comfortable and precise imaging process. The digital impressions are then utilized to design and fabricate maxillary dentures using 3D printing technology. The intervention focuses on evaluating patient satisfaction with the dentures in terms of comfort, fit, and aesthetics.
Device: Extra orally scanned — The extra-oral scanning method involves creating conventional impressions of the oral cavity using traditional impression materials. These impressions are then scanned externally using the 3Shape scanner to produce digital models. The digital models are used to design and fabricate maxillary dentures through 3D printing technology. This intervention aims to assess patient satisfaction with the dentures based on comfort, fit, and aesthetics.

SUMMARY:
The goal of this clinical trial is to evaluate patient satisfaction with intra-orally scanned versus extra-orally scanned digitally printed maxillary dentures in completely edentulous patients. The main questions it aims to answer are:

1. Do intra-orally scanned dentures provide higher patient satisfaction compared to extra-orally scanned dentures?
2. Are there significant differences in comfort, fit, aesthetics and phonetics between the two types of dentures?

Researchers will compare the intra-orally scanned denture group to the extra-orally scanned denture group to determine if one method leads to superior patient-reported outcomes.

Participants will:

* Receive both types of dentures (intra-orally scanned and extra-orally scanned), with a three-week wash-out period between each intervention.
* Complete satisfaction surveys to assess comfort, fit, and aesthetics after using each type of denture.

The study aims to provide evidence on the optimal scanning method for digitally printed maxillary dentures in edentulous patients.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate and compare patient satisfaction with intra-orally scanned and extra-orally scanned digitally printed maxillary dentures in completely edentulous patients. This in vivo study seeks to provide insights into how the scanning method impacts the comfort, fit, and aesthetics of maxillary dentures, ultimately guiding clinicians in choosing the most patient-preferred approach.

Study Design and Objectives

This study involves eight completely edentulous participants who will receive both types of dentures-one set based on intra-oral scanning and another based on extra-oral scanning. A wash-out period of two weeks between the use of each denture ensures that the effects of one intervention do not influence the results of the other. The primary objectives of this study are:

1. To determine if intra-orally scanned dentures provide higher patient satisfaction compared to extra-orally scanned dentures.
2. To assess specific satisfaction factors, including comfort, fit, and aesthetic appearance, for both denture types.

Study Methodology

Participants will undergo the following steps:

1. Scans and Fabrication:

   * Intra-oral scanning will be performed using the 3Shape scanner to capture precise digital impressions of the oral cavity.
   * For the extra-oral scanning, conventional impressions will first be taken, and these will be scanned externally using the same scanner to create digital models.
   * Both types of digital models will be used to fabricate maxillary dentures using 3D printing technology.
2. Fitting and Wash-out Period:

   * Participants will first use one type of denture (either intra-oral or extra-oral scanned) for a designated period.
   * After a two-week wash-out period without wearing dentures, they will switch to the other type of denture.
3. Data Collection:

   * After wearing each type of denture, participants will complete structured satisfaction questionnaire focusing on key parameters: comfort during daily use, overall fit, and aesthetic appeal.

Data Analysis

The study will compare satisfaction scores and qualitative responses between the two scanning methods. Statistical analyses will be conducted to identify significant differences in patient-reported outcomes.

Expected Impact

This study aims to provide clinicians with evidence-based guidance on whether intra-oral or extra-oral scanning results in better patient satisfaction for digitally printed maxillary dentures. By focusing on the user experience, this research contributes to improving prosthodontic care for completely edentulous patients.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients
* Angle's Class I skeletal relationship
* Normal facial symmetry
* Cooperative patients

Exclusion Criteria:

* -Temporomandibular disorders
* Uncontrolled diabetes
* Patient's with neuromuscular disorders
* Severe psychiatric disorders
* Angle's class II and III skeletal relationship.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-12-03 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | Assessment will be conducted after patient delivery at 6 months after wearing each denture where as a washout period of two weeks will be observed between the two interventions.
  Patient satisfaction will be assessed using a Visual Analogue Scale questionnaire covering cleanliness, comfort, esthetics,phonetics and fit

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry-Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No